CLINICAL TRIAL: NCT02196714
Title: A Phase I, Randomized, Double-Blind, Single-Dose, Four-Period, Four-Treatment, Cross-Over Study Evaluating the Safety and Pharmacokinetics of Two Doses of PT003 and Two Doses of PT001 in Japanese Healthy Subjects
Brief Title: PK Study of PT003 and PT001 in Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PT003010-00
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: COPD
Keywords: Japanese Healthy Volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glycopyrronium and Formoterol Fumarate (GFF) Dose 1 (Experimental): Glycopyrronium and Formoterol Fumarate metered-dose inhaler MDI (GFF MDI), Dose 1; PT003 administered as 2 inhalations twice-daily (BID)
  Interventions: Drug: Glycopyrronium and Formoterol Fumarate (GFF) Dose 1
- Glycopyrronium and Formoterol Fumarate (GFF) Dose 2 (Experimental): Glycopyrronium and Formoterol Fumarate metered-dose inhaler MDI (GFF MDI), Dose 2; PT003 administered as 2 inhalations twice-daily (BID)
  Interventions: Drug: Glycopyrronium and Formoterol Fumarate (GFF) Dose 2
- Glycopyrronium (GP) Dose 1 (Experimental): Glycopyrronium metered-dose inhaler MDI (GP MDI), Dose 1; PT001 administered as 2 inhalations twice-daily (BID)
  Interventions: Drug: Glycopyrronium (GP) Dose 1
- Glycopyrronium (GP) Dose 2 (Experimental): Glycopyrronium metered-dose inhaler MDI (GP MDI), Dose 2; PT001 administered as 2 inhalations twice-daily (BID)
  Interventions: Drug: Glycopyrronium (GP) Dose 2

INTERVENTIONS:
Drug: Glycopyrronium and Formoterol Fumarate (GFF) Dose 1 — Glycopyrronium and Formoterol Fumarate metered-dose inhaler MDI (GFF MDI), Dose 1; PT003 administered as 2 inhalations twice-daily (BID)
  Arms: Glycopyrronium and Formoterol Fumarate (GFF) Dose 1
Drug: Glycopyrronium and Formoterol Fumarate (GFF) Dose 2 — Glycopyrronium and Formoterol Fumarate metered-dose inhaler MDI (GFF MDI), Dose 2; PT003 administered as 2 inhalations twice-daily (BID)
  Arms: Glycopyrronium and Formoterol Fumarate (GFF) Dose 2
Drug: Glycopyrronium (GP) Dose 1 — Glycopyrronium metered-dose inhaler MDI (GP MDI), Dose 1; PT001 administered as 2 inhalations twice-daily (BID)
  Arms: Glycopyrronium (GP) Dose 1
Drug: Glycopyrronium (GP) Dose 2 — Glycopyrronium metered-dose inhaler MDI (GP MDI), Dose 2; PT001 administered as 2 inhalations twice-daily (BID)
  Arms: Glycopyrronium (GP) Dose 2

SUMMARY:
A Randomized, Double-Blind, Single-Dose, Four-Period, Four-Treatment, Cross-Over, Single-Center, Phase I, Crossover Study in Healthy Japanese Adult Subjects to Evaluate the Safety and Pharmacokinetics of Two Doses of PT003 and Two Doses of PT001.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent Form (ICF) prior to any study related procedures

* Male and female first generation Japanese subjects 18 to 45 years, inclusive
* Good general health
* Medically acceptable contraception for women of child-bearing potential and males with female partners of childbearing potential
* Clinical labs within normal ranges or determined to be not clinically significant by the Investigator

Exclusion Criteria:

* Pregnancy, nursing female subjects, or subjects trying to conceive
* Clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematological, psychiatric, or other medical illness that would interfere with participation in this study
* History of ECG abnormalities
* Cancer not in complete remission for at least 5 years
* Clinically significant, symptomatic prostatic hypertrophy
* Male subjects with a trans-urethral resection of the prostate or full resection of the prostate within 6 months prior to Screening
* Clinically significant bladder neck obstruction or urinary retention
* Inadequately treated glaucoma
* History of an allergic reaction or hypersensitivity to any drug or to any component of the formulations used in this study
* Subjects with pre-existing anemia and/or iron deficiency

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Orevillo, Study Chair — Pearl Therapeutics, Inc.
Locations (1):
- SNBL, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Reisner C, Miller J, DePetrillo P, Maes A, Siddiqui S, Martin UJ. Pharmacokinetics and safety of a single dose of the novel LAMA/LABA fixed-dose combination of glycopyrronium/formoterol fumarate dihydrate metered dose inhaler, formulated using co-suspension delivery technology, in Japanese healthy subjects. Pulm Pharmacol Ther. 2018 Dec;53:33-38. doi: 10.1016/j.pupt.2018.09.005. Epub 2018 Sep 13. PMID 30218695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 1 site from July 2014 - September 2014. Study duration for each subject was between 33 and 98 days.
Pre-assignment Details: Study was four-period, four-treatment, complete cross-over design in healthy adult Japanese Subjects. Each treatment visit was followed by a minimum 7 day to maximum 14 day washout period between treatments.
Groups:
- Received GFF MDI 28.8/9.6 μg: Glycopyrronium and Formoterol Fumurate (GFF) Metered Dose Inhaler (MDI) 28.8/9.6 μg
- Received GFF MDI 14.4/9.6 μg: Received GFF MDI 14.4/9.6 μg
- Received GP MDI 28.8 μg: Glycopyrronium (GP) Metered Dose Inhaler (MDI) 28.8 μg
- Received GP MDI 14.4 μg: Received GP MDI 14.4 μg
Period: Overall Study
Arm/Group | Received GFF MDI 28.8/9.6 μg | Received GFF MDI 14.4/9.6 μg | Received GP MDI 28.8 μg | Received GP MDI 14.4 μg
Started | 24 | 23 | 24 | 24
Completed | 24 | 23 | 23 | 24
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis Set: All Subjects Randomized
Groups:
- All Subjects: Analysis Set: All Subjects Randomized
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment (Cmax)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: pg/mL
Groups:
- GFF MDI 28.8/9.6 ug: Glycopyrronium and Formoterol Fumurate (GFF) Metered Dose Inhaler (MDI) 28.8/9.6 ug
- GFF MDI 14.4/9.6 ug: GFF MDI 14.4/9.6 ug
- GP MDI 28.8 ug: GP MDI 28.8 ug
- GP MDI 14.4 µg: GP MDI 14.4 µg
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug | GP MDI 14.4 µg
Number analyzed (Participants) | 24 | 22 | 24 | 23
pg/mL | 15.23 (7.69) [2.11 to 38.80] | 9.09 (6.5) [2.25 to 27.80] | 16.85 (4.26) [4.09 to 56.40] | 7.26 [2.51 to 16.10]

2. Primary Outcome: Cmax
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment (Cmax)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 24 | 23
pg/mL | 10.74 (3.46) [3.18 to 16.20] | 11.99 (7.07) [3.95 to 30.90]

3. Primary Outcome: AUC 0-12
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment (AUC 0-12)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: h*pg/mL
Groups:
- GP MDI 14.4 ug: GP MDI 14.4 ug
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug | GP MDI 14.4 ug
Number analyzed (Participants) | 24 | 22 | 24 | 23
h*pg/mL | 45.43 (19.43) [11.31 to 83.76] | 21.75 (9.00) [3.71 to 43.16] | 50.59 (10.75) [13.57 to 108.54] | 24.72 [7.63 to 51.06]

4. Primary Outcome: AUC 0-12
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment (AUC 0-12)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: h*pg/mL
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 24 | 23
h*pg/mL | 44.15 (15.3) [10.59 to 79.35] | 42.54 (12.04) [17.88 to 62.21]

5. Primary Outcome: AUC 0-t
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment (AUC 0-t)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: h*pg/mL
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug | GP MDI 14.4 µg
Number analyzed (Participants) | 24 | 22 | 24 | 23
h*pg/mL | 53.52 (3.31) [7.11 to 122.09] | 21.37 (14.53) [1.49 to 58.08] | 64.05 (17.61) [9.69 to 146.37] | 23.72 [5.27 to 68.02]

6. Primary Outcome: AUC 0-t
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment (AUC 0-t)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: h*pg/mL
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 24 | 23
h*pg/mL | 45.96 (19.85) [7.94 to 107.41] | 42.39 (14.69) [14.93 to 69.75]

7. Primary Outcome: AUC 0-∞
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment (AUC 0-∞)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: h*pg/mL
Groups:
- GP MDI 28.8 µg: GP MDI 28.8 µg
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 µg | GP MDI 14.4 µg
Number analyzed (Participants) | 7 | 2 | 2 | 3
h*pg/mL | 46.26 [29.58 to 60.11] | 32.18 [30.24 to 34.13] | 37.32 [32.36 to 42.28] | 34.04 [33.67 to 34.64]

8. Primary Outcome: AUC 0-∞
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment (AUC 0-∞)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: h*pg/mL
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 16 | 11
h*pg/mL | 61.88 (21.60) [41.27 to 126.07] | 61.43 (12.01) [45.43 to 82.84]

9. Primary Outcome: Tmax
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment (tmax)
Time Frame: Day 1
Population: Pharmacokinetic Population
Measure: Mean (Full Range); unit: h
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug | GP MDI 14.4 ug
Number analyzed (Participants) | 24 | 22 | 24 | 23
h | 0.10 [0.03 to 4.02] | 0.10 [0.03 to 0.10] | 0.10 [0.03 to 2.00] | 0.10 [0.03 to 4.10]

10. Primary Outcome: Tmax
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment (tmax)
Time Frame: Day 1
Population: Pharmacokinetic Population
Measure: Mean (Full Range); unit: h
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 24 | 23
h | 0.10 [0.10 to 1.00] | 0.10 [0.10 to 2.00]

11. Primary Outcome: T 1/2
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment (T 1/2)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: h
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug | GP MDI 14.4 ug
Number analyzed (Participants) | 14 | 14 | 10 | 13
h | 9.49 (11.98) [2.88 to 37.90] | 4.14 (1.40) [1.31 to 6.89] | 24.87 (51.77) [2.14 to 103.21] | 19.13 [2.08 to 191.29]

12. Primary Outcome: T 1/2
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment (T 1/2)
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: h
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 21 | 20
h | 5.45 (2.39) [3.11 to 14.36] | 5.25 (2.32) [3.24 to 13.87]

13. Primary Outcome: CL/F
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: L/h
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 µg | GP MDI 14.4 µg
Number analyzed (Participants) | 7 | 2 | 2 | 3
L/h | 657.91 [479.15 to 973.62] | 449.10 [421.97 to 476.24] | 785.60 [681.20 to 890.00] | 423.12 [415.74 to 427.70]

14. Primary Outcome: CL/F
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: L/h
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 7 | 2
L/h | 168.95 (45.28) [76.15 to 232.63] | 161.55 (30.17) [151.89 to 211.32]

15. Primary Outcome: Vd/F
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrroniuml by Treatment
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 µg | GP MDI 14.4 µg
Number analyzed (Participants) | 7 | 2 | 2 | 3
L | 3508.00 [2089.69 to 4654.28] | 2577.78 [2475.12 to 2680.44] | 3555.88 [3509.62 to 3602.14] | 2101.03 [1929.07 to 2193.02]

16. Primary Outcome: Vd/F
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 7 | 2
L | 1187.75 (313.20) [516.40 to 1779.88] | 1054.16 (225.15) [828.09 to 1618.22]

17. Primary Outcome: Lambda z
Description: Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: 1/h
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug | GP MDI 14.4 ug
Number analyzed (Participants) | 14 | 14 | 10 | 13
1/h | 0.1506 (7.69) [0.0183 to 0.2404] | 0.1983 (6.5) [0.1007 to 0.5299] | 0.1100 (4.26) [0.0067 to 0.3242] | 0.1614 [0.0036 to 0.3333]

18. Primary Outcome: Lambda z
Description: Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment
Time Frame: Day 1
Population: Pharmacokinetic Population (includes subjects with an evaluable profile for this analyte)
Measure: Mean (Full Range); unit: 1/h
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug
Number analyzed (Participants) | 14 | 14
1/h | 0.1412 (0.0381) [0.0483 to 0.2225] | 0.1470 (0.0410) [0.0500 to 0.2140]

19. Secondary Outcome: Change in Mean Hematology Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose
Time Frame: 12 Hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9cells/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
10^9cells/L
  Basophils (10^9cells/L) | 0.007 (0.025) | 0.000 (0.022) | 0.001 (0.028)
  Eosinophils (10^9cells/L) | 0.044 (0.048) | 0.033 (0.068) | 0.065 (0.103)
  Granulocytes (10^9cells/L) | 0.222 (1.436) | 0.483 (1.793) | 0.443 (1.278)
  Leukocytes (10^9cells/L) | 0.484 (1.710) | 0.780 (1.990) | 0.800 (1.526)
  Lymphocytes (10^9cells/L) | 0.147 (0.390) | 0.206 (0.402) | 0.235 (0.383)
  Monocytes (10^9cells/L) | 0.065 (0.084) | 0.056 (0.115) | 0.055 (0.103)
  Platelets (10^9cells/L) | -22.4 (24.5) | -14.4 (16.2) | -23.1 (26.6)

20. Secondary Outcome: Change in Mean Hematology Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose
Time Frame: 12 Hours
Description (as registered): Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose (Ery. mean corpuscuar volume)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
Ratio
  Basophils/leukocytes (ratio) | -0.0001 (0.0044) | -0.0013 (0.0040) | -0.0013 (0.0039)
  Eosinophils/leukocytes (ratio) | 0.0034 (0.0089) | 0.0026 (0.0131) | 0.0046 (0.0091)
  Granulocytes/leukocytes (ratio) | 0.0043 (0.0688) | 0.0003 (0.0818) | -0.0010 (0.0759)
  Hematocrit (ratio) | -0.040 (0.022) | -0.041 (0.030) | -0.043 (0.023)
  Lymphocytes/leukocytes (ratio) | -0.0110 (0.0565) | -0.0019 (0.0662) | -0.0018 (0.0616)
  Monocytes/leukocytes (ratio) | 0.0034 (0.0125) | 0.0004 (0.0136) | -0.0006 (0.0118)

21. Secondary Outcome: Change in Mean Hematology Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose
Time Frame: 12 Hours
Description (as registered): Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose (Ery. mean corpuscuar hemoglobin)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
g/L
  Ery. mean corpuscuar HGB (g/L) | 12.0 (15.5) | 8.5 (13.9) | 11.4 (15.2)
  Hemoglobin (g/L) | -8.81 (7.76) | -10.61 (9.10) | -10.38 (9.10)

22. Secondary Outcome: Change in Mean Hematology Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose (Ery. mean corpuscuar volume)
Time Frame: 12 Hours
Description (as registered): Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose (Erythrocytes)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
fL | -0.9 (0.6) | -0.8 (0.9) | -0.9 (0.8)

23. Secondary Outcome: Change in Mean Hematology Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose (Ery. mean corpuscuar hemoglobin)
Time Frame: 12 Hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pg/cell
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
pg/cell | 0.78 (1.29) | 0.49 (1.08) | 0.75 (1.22)

24. Secondary Outcome: Change in Mean Hematology Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Hematology Parameters (±SD) from Pre-dose to 12 Hours Post-dose (Erythrocytes)
Time Frame: 12 Hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12cells/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
10^12cells/L | -0.391 (0.242) | -0.419 (0.326) | -0.433 (0.253)

25. Secondary Outcome: Change in Mean Chemistry Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Chemistry Parameters (±SD) from Pre-dose to 12 Hours Post-dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
IU/L
  ALT (IU/L) | -3.1 (4.3) | -1.7 (3.1) | -2.4 (3.9)
  Alkaline phosphatase (IU/L) | -5.2 (4.3) | -5.0 (5.1) | -6.0 (3.1)
  AST (IU/L) | -4.2 (3.7) | -3.3 (2.6) | -3.7 (3.0)
  Gamma glutamyl transferase (IU/L) | -2.5 (2.4) | -1.6 (1.9) | -2.2 (1.9)

26. Secondary Outcome: Change in Mean Chemistry Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Chemistry Parameters (±SD) from Pre-dose to 12 Hours Post-dose
Time Frame: 12 hours
Description (as registered): Change in Mean Chemistry Parameters (±SD) from Pre-dose to 12 Hours Post-dose (eGFR)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
g/L
  Albumin (g/L) | -7.1 (2.9) | -6.9 (4.1) | -6.7 (2.4)
  Protein (g/L) | -10.9 (5.3) | -10.8 (6.7) | -10.3 (4.3)

27. Secondary Outcome: Change in Mean Chemistry Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Chemistry Parameters (±SD) from Pre-dose to 12 Hours Post-dose
Time Frame: 12 hours
Description (as registered): Change in Mean Chemistry Parameters (±SD) from Pre-dose to 12 Hours Post-dose (Ferritin)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
mmol/L
  Blood urea nitrogen (mmol/L) | 0.01 (1.45) | 0.34 (1.32) | 0.74 (1.51)
  Calcium (mmol/L) | -0.15 (0.09) | -0.14 (0.12) | -0.13 (0.06)
  Chloride (mmol/L) | 3.0 (2.3) | 2.5 (1.8) | 2.3 (1.5)
  Magnesium (mmol/L) | -0.05 (0.09) | -0.07 (0.09) | -0.04 (0.20)
  Phosphorus (mmol/L) | 0.135 (0.165) | 0.163 (0.132) | 0.133 (0.164)
  Sodium (mmol/L) | 0.9 (2.1) | 0.5 (1.3) | 0.1 (1.6)

28. Secondary Outcome: Change in Mean Chemistry Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Chemistry Parameters (±SD) from Pre-dose to 12 Hours Post-dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
μmol/L
  Creatinine (μmol/L) | 1.88 (11.14) | 4.92 (15.74) | 3.61 (13.41)
  Direct bilirubin (μmol/L) | -3.06 (1.75) | -2.53 (1.45) | -2.64 (2.14)
  Iron (μmol/L) | -5.42524 (8.9) | -2.81888 (7.07702) | -2.58949 (8.19974)
  Total bilirubin (μmol/L) | -8.19 (5.68) | -7.14 (4.80) | -7.20 (5.92)

29. Secondary Outcome: Change in Mean Chemistry Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Chemistry Parameters (±SD) from Pre-dose to 12 Hours Post-dose (eGFR)
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
mL/min/1.73m2 | -4.2 (13.2) | -7.2 (16.6) | -3.5 (15.3)

30. Secondary Outcome: Change in Mean Chemistry Parameters (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Chemistry Parameters (±SD) from Pre-dose to 12 Hours Post-dose (Ferritin)
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
μg/L | -14.169 (13.912) | -11.949 (12.306) | -11.669 (9.731)

31. Secondary Outcome: Change in Mean Glucose and Potassium Results (±SD) From Pre-dose to 12 Hours Post-dose
Description: Change in Mean Glucose and Potassium Results (±SD) from Pre-dose to 12 Hours Post-dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
mmol/L
  Glucose (mmol/L) 30 minutes post-dose | -0.03 [-0.3 to 0.6] | -0.08 [-0.8 to 0.5] | -0.01 [-0.4 to 0.7]
  Glucose (mmol/L) 2 hours post-dose | 0.05 [-0.3 to 0.4] | -0.01 [-0.7 to 0.8] | -0.06 [-0.4 to 0.7]
  Glucose (mmol/L) 4 hours post-dose | -0.08 [-0.5 to 0.4] | -0.24 [-0.8 to 0.4] | -0.16 [-0.6 to 0.7]
  Glucose (mmol/L) 12 hours post-dose | 0.10 [-0.4 to 0.7] | 0.18 [-0.8 to 0.8] | 0.23 [-0.3 to 0.9]
  Potassium (mmol/L) 30 minutes post-dose | 0.01 [-0.3 to 1.0] | 0.00 [-0.6 to 0.5] | 0.06 [-0.5 to 0.9]
  Potassium (mmol/L) 2 hours post-dose | -0.02 [-0.5 to 0.8] | -0.07 [-0.5 to 0.4] | 0.10 [-0.4 to 2.4]
  Potassium (mmol/L) 4 hours post-dose | -0.01 [-0.6 to 1.0] | -0.12 [-0.5 to 0.4] | -0.07 [-0.6 to 0.4]
  Potassium (mmol/L) 12 hours post-dose | 0.05 [-0.5 to 0.7] | -0.06 [-0.6 to 0.4] | 0.07 [-0.5 to 1.0]

32. Secondary Outcome: Change in Heart Rate From Pre-dose to 12 Hours Post Dose
Description: Change in Heart Rate from Pre-dose to 12 hours Post dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Full Range); unit: Beats/Min
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
Beats/Min | 11.3 [2 to 42] | 9.3 [-4 to 36] | 4.5 [-13 to 29]

33. Secondary Outcome: Change in PR Interval From Pre-dose to 12 Hours Post Dose
Description: Change in PR Interval from Pre-dose to 12 hours Post dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Full Range); unit: msec
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
msec | -10.7 [-22 to 6] | -8.5 [-46 to 14] | -7.4 [-36 to 6]

34. Secondary Outcome: Change in QRS Axis From Pre-dose to 12 Hours Post Dose
Description: Change in QRS axis from Pre-dose to 12 hours Post dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Full Range); unit: QRS axis
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
QRS axis | -0.5 [-20 to 15] | 4.1 [-11 to 76] | 0.0 [-21 to 16]

35. Secondary Outcome: Change in QRS Duration From Pre-dose to 12 Hours Post Dose
Description: Change in QRS duration from Pre-dose to 12 hours Post dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Full Range); unit: msec
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
msec | -3.9 [-24 to 8] | -1.1 [-14 to 6] | -4.0 [-22 to 4]

36. Secondary Outcome: Change in QT Interval From Pre-dose to 12 Hours Post Dose
Description: Change in QT Interval from Pre-dose to 12 hours Post dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Full Range); unit: msec
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
msec | -28.5 [-64 to 0] | -24.8 [-78 to 0] | -20.5 [-72 to 24]

37. Secondary Outcome: Change in QTc Bazett Interval From Pre-dose to 12 Hours Post Dose
Description: Change in QTc Bazett Interval from Pre-dose to 12 hours Post dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Full Range); unit: msec
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
msec | 7.2 [-14 to 40] | 4.4 [-26 to 30] | -5.8 [-28 to 10]

38. Secondary Outcome: Change in QTc Fridericia's Interval From Pre-dose to 12 Hours Post Dose
Description: Change in QTc Fridericia's Interval from Pre-dose to 12 hours Post dose
Time Frame: 12 hours
Population: Safety Population
Measure: Mean (Full Range); unit: msec
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug
Number analyzed (Participants) | 24 | 23 | 24
msec | -4.8 [-17 to 11] | -5.4 [-27 to 16] | -10.8 [-29 to 5]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Day 0 (Randomization visit and first dose) through Final Follow-up Visit, which is 7-14 days post final dose.
Description: Serious Adverse Events collected from time subject signs ICF, up to 14 days following the last dose of study drug.
Arm/Group | GFF MDI 28.8/9.6 ug | GFF MDI 14.4/9.6 ug | GP MDI 28.8 ug | GP MDI 14.4 µg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 8/23 | 4/24 | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI 28.8/9.6 ug (N=24) | GFF MDI 14.4/9.6 ug (N=23) | GP MDI 28.8 ug (N=24) | GP MDI 14.4 µg (N=24)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.